CLINICAL TRIAL: NCT05413421
Title: An Open-Label, Phase 1/1b Study of ORIC-944 as a Single Agent or in Combination With an Androgen Receptor Pathway Inhibitor in Patients With Metastatic Prostate Cancer
Brief Title: Study of ORIC-944 in Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-944-01
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: PRC2 dysregulation; EED; CRPC; mCRPC; ARPI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; darolutamide; enzalutamide

STUDY DESIGN:
Intervention Model Description: Interval 3+3 dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Agent Dose Escalation (Experimental): ORIC-944 dosed orally on a continuous daily dosing regimen in 28-day cycles
  Interventions: Drug: ORIC-944
- Combination Dose Escalation (Experimental): ORIC-944 dosed orally on a continuous daily dosing regimen in 28-day cycles in combinations with abiraterone, apalutamide, darolutamide, or enzalutamide
  Interventions: Drug: ORIC-944; Drug: Abiraterone acetate (Zytiga®) 250 mg or 500 mg tablets; Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets; Drug: Darolutamide (Nubeqa®) 300 mg tablets; Drug: Enzalutamide (Xtandi®) 40 mg capsules or 40 mg and 80 mg tablets
- Combination Dose Optimization (Experimental): Cohort A and C: ORIC-944 dosed orally on a continuous daily dosing regimen in 28-day cycles in combination with apalutamide
  Cohort B and D: ORIC-944 dosed orally on a continuous daily dosing regimen in 28-day cycles in combination with darolutamide
  Combinations with abiraterone or enzalutamide may be conducted in the future
  Interventions: Drug: ORIC-944; Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets; Drug: Darolutamide (Nubeqa®) 300 mg tablets

INTERVENTIONS:
Drug: ORIC-944 — Oral, once daily, continuous
Drug: Abiraterone acetate (Zytiga®) 250 mg or 500 mg tablets — Oral, 1000 mg once daily, continuous
  Arms: Combination Dose Escalation
Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets — Oral, 240 mg once daily, continuous
  Arms: Combination Dose Escalation; Combination Dose Optimization
Drug: Darolutamide (Nubeqa®) 300 mg tablets — Oral, 600 mg twice daily, continuous
  Arms: Combination Dose Escalation; Combination Dose Optimization
Drug: Enzalutamide (Xtandi®) 40 mg capsules or 40 mg and 80 mg tablets — Oral, 160 mg once daily, continuous
  Arms: Combination Dose Escalation

SUMMARY:
The purpose of this study is to establish the safety and preliminary antitumor activity of ORIC-944 as a single agent and in combinations with ARPIs in patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
ORIC-944 is a potent, highly selective, allosteric, orally bioavailable, small molecule inhibitor of PRC2 via binding the embryonic ectoderm development (EED) subunit.

This is a first-in-human, open-label, multicenter, dose escalation study of ORIC-944 as a single agent (Part I) or in combination with an Androgen Receptor Pathway Inhibitor (ARPI) (Part II) to establish the safety and preliminary antitumor activity of ORIC-944 as a single agent and in combination with ARPIs in patients with metastatic prostate cancer. Part III of the protocol (dose optimization) will explore two potential dose levels of ORIC-944 selected from Part II in combination with ARPIs to select the final RP2D for each combination across two separate patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic prostate cancer
* Must have undergone bilateral orchiectomy or be willing to continue GnRH analogue or antagonist to maintain castrate levels of testosterone
* Prior therapies:

Part I (single agent ORIC-944 dose escalation): Any number of prior therapies are allowed, but must have progressed after at least one line of next generation ARPI (abiraterone, apalutamide, darolutamide, or enzalutamide) and must not have received more than 2 chemotherapy regimens in the mCRPC setting

Part II (ARPI combination dose escalation): Must have received only 1 prior line of ARPI (abiraterone, apalutamide, darolutamide, or enzalutamide) in any setting; may have also received up to 1 prior line of chemotherapy in the mCSPC setting

Part III (ARPI combination dose optimization): In addition to up to 1 prior line of chemotherapy in the mCSPC setting:

* Cohorts A and B: received only one 1 prior line of abiraterone in any setting
* Cohorts C and D: received only one 1 prior line of apalutamide, darolutamide, or enzalutamide in any setting:

  * Evidence of progressive disease by PCWG3 criteria for study entry

    * rising PSA, defined as a minimum of 2 rising values obtained a minimum of one week apart with the latest result being at least 2.0 ng/mL (or 1.0 ng/mL if PSA rise is the only indication of progression), or
    * confirmation of 2 new bone lesions on last systemic therapy, or
    * soft tissue progression per RECIST 1.1
  * Measurable and/or evaluable disease by RECIST 1.1
  * Agreement and ability to undergo on-study punch skin biopsies and core tumor biopsies
  * ECOG performance status of 0 or 1
  * Adequate organ function

Exclusion Criteria:

* History or presence of CNS metastases, unless previously treated and stable
* History of class III or IV congestive heart failure or severe non-ischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months
* Known, symptomatic human immunodeficiency virus (HIV) infection
* Active symptomatic Hepatitis B or C infection; patients with well controlled disease are eligible
* Active gastrointestinal disease (eg, Crohn's disease, ulcerative colitis, short gut syndrome, etc) or other malabsorption syndromes that would reasonably impact drug absorption per investigator judgement
* Any other condition or circumstance (eg, clinical, psychological, familial, sociological, inability to swallow oral study drug) that, in the opinion of the investigator, may interfere with protocol compliance or contraindicates participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D as determined by interval 3+3 dose escalation design
Maximum plasma concentration (Cmax) | 28 Days
  PK of ORIC-944 single agent and in combination with an ARPI
Time to maximum observed concentration (Tmax) | 28 Days
  PK of ORIC-944 single agent and in combination with an ARPI
Area under the curve (AUC) | 28 Days
  PK of ORIC-944 single agent and in combination with an ARPI
Apparent plasma terminal elimination half-life (t1/2) | 28 Days
  PK of ORIC-944 single agent and in combination with an ARPI

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Objective response rate (ORR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response (DOR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-free survival (PFS) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
On-treatment PSA levels and change from baseline | 36 months
  Prostate cancer working group 3 criteria (PCWG3)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, Study Director — ORIC Pharmaceuticals
Locations (27):
- United States (20):
  - Rocky Mountain Cancer Center, Colorado Springs, Colorado
  - South Florida Oncology and Hematology, Plantation, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - First Urology, Jeffersonville, Indiana
  - Marlene & Stewart Greenebaum Comprehensive Cancer Center, University of Maryland, Baltimore, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Karmanos, Detroit, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Memorial Sloane Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Amarillo Urology Research, Amarillo, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Oncology Associates, Fairfax, Virginia
  - Virginia Cancer Specialists, Norfolk, Virginia
  - University of Washington, Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (3):
  - Sydney Adventist Health, Wahroonga, New South Wales
  - Bendigo Health, Bendigo, Victoria
  - Peninsula Health, Frankston, Victoria
- Spain (3):
  - NEXT Oncology, Barcelona, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona, Barcelona
  - NEXT Oncology, Madrid
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom